CLINICAL TRIAL: NCT05105152
Title: Pediatric And Young Adult Leukemia Adoptive Therapy (PLAT)-08: A Phase 1 Study Of SC-DARIC33 In Pediatric And Young Adults With Relapsed Or Refractory CD33+ AML
Brief Title: PLAT-08: A Study Of SC-DARIC33 CAR T Cells In Pediatric And Young Adults With Relapsed Or Refractory CD33+ AML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Colleen Annesley, Medical Director, Seattle Children's Therapeutics, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLAT-08
Record Dates: First submitted 2021-10-07; First posted 2021-11-03 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia Refractory; Acute Myeloid Leukemia, in Relapse
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Phase I open-label, dose-finding study employing the Bayesian optimal interval (BOIN) design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DARIC-33 (Experimental)
  Interventions: Biological: SC-DARIC33

INTERVENTIONS:
Biological: SC-DARIC33 — Infusion with SC-DARIC33 followed by intermittent oral rapamycin administration

SUMMARY:
A phase 1, open-label, non-randomized study enrolling pediatric and young adult patients with relapsed or refractory CD33+ leukemia with and without prior history of allogeneic hematopoietic cell transplantation, to examine the safety and feasibility of administering an autologous T cell product that has been genetically modified to express a Dimerizing Agent Regulated Immunoreceptor Complex (DARIC).

ELIGIBILITY:
Inclusion Criteria:

1. Subject age ≤ 30 years. The first three enrolled subjects must be ≥ 18 years of age.
2. AML that expresses CD33 by flow cytometry and meets one of the below definitions:

   1. For subjects who have previously received an allogeneic HCT, any evidence of AML re-emergence post HCT detectable by flow cytometry
   2. First relapse of AML ≤ 6 months of initial diagnosis
   3. First relapse of AML > 6 months after initial diagnosis, with MRD of >0.1% by flow cytometry (MPF) after at least one re-induction (single cycle) attempt
   4. Second or greater relapse AML
   5. Refractory AML, defined as >1% leukemic cells determined by flow cytometry after 2 cycles of induction chemotherapy
3. Able to tolerate apheresis, or subject with sufficient existing apheresis product or T cells for manufacturing investigational product.
4. Life expectancy ≥ 8 weeks
5. Has an appropriate stem cell donor source identified
6. Lansky performance status score of ≥ 50 for subjects <16 years of age or Karnofsky score ≥ 50 for subjects ≥ 16 years. Subjects who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for purposes of assessing performance status
7. If a subject does not have a previously obtained apheresis product that is acceptable and available for manufacturing of DARIC T cells, the subject must discontinue all anticancer agents and radiotherapy and, in the opinion of the investigator, have fully recovered from significant acute toxic effects of all prior chemotherapy, immunotherapy, and radiotherapy:

   a. Chemotherapy and biologic agents: All chemotherapy and biologic therapy not specifically mentioned below must be discontinued ≥ 7 days prior to enrollment, with the exception of intrathecal chemotherapy for which there is not a required washout period b. Must be ≥ 30 days from last gemtuzumab ozogamicin dose. c. Steroid use: All corticosteroid therapy (unless physiologic replacement dosing) must be discontinued ≥ 7 days prior to enrollment d. Tyrosine Kinase Inhibitor (TKI) use: All TKIs must be discontinued ≥ 3 days prior to enrollment e. Hydroxyurea: must be discontinued ≥ 1 day prior to enrollment. f. Gene Modified cellular therapy: i. must be at least 30 days from most recent gene modified cell therapy infusion and document no evidence of modified cells in the peripheral blood OR ii. must be at least 60 days from most recent gene modified cell therapy
8. Adequate organ function as indicated by:

   1. Renal: Serum creatinine ≤ 1.5 X the upper limit of normal (ULN)
   2. Hepatic: Total bilirubin ≤ 3 times ULN for age OR conjugated bilirubin ≤ 2 mg/dL AND ALT (SGPT) ≤ 5 times ULN
   3. Cardiac: Shortening fraction ≥ 28% OR ejection fraction ≥ 50% as measured by echocardiogram
   4. Respiratory: Oxygen saturation ≥ 92% on room air without supplemental oxygen or mechanical ventilation
9. Laboratory values meet the following criteria:

   a. Subjects requiring apheresis: Absolute Lymphocyte Count (ALC) ≥ 100 cells/uL b. Virology Testing negative within 3 months prior to enrollment, to include: i. HIV antigen & antibody ii. Hepatitis B surface antigen iii. Hepatitis C antibody OR if positive, Hepatitis C PCR is negative
10. If subject is of childbearing or child-fathering potential, must agree to use highly effective contraception from the time of initial consent through 12 months following the infusion of investigational product on this trial.
11. Subject and/or legally authorized representative has signed the Informed Consent Form for this study

Exclusion Criteria:

1. Active malignancy other than acute myeloid leukemia
2. History of symptomatic non-AML CNS disease or ongoing symptomatic CNS disease requiring medical intervention, including paresis, aphasia, cerebrovascular ischemia/hemorrhage, severe brain injury, dementia, cerebellar disease, organic brain syndrome, psychosis, coordination or movement disorder (subjects with non-febrile seizure disorder controlled on anti-epileptic medication and without seizure activity within 1 month are eligible).
3. CNS AML involvement that is symptomatic and in the opinion of the investigator, cannot be controlled during the interval between enrollment and DARIC T cell infusion
4. If history of allogeneic stem cell transplant: active GVHD, or receiving immunosuppressive therapy for treatment or prevention of GVHD within 4 weeks prior to enrollment
5. Presence of active severe infection, defined as:

   i. positive blood culture within 48 hours of enrollment, OR ii. fever above 38.2° C, AND clinical signs of infection within 48 hours of enrollment
6. Primary immunodeficiency syndrome
7. Subject has received prior virotherapy
8. Pregnant or breastfeeding
9. Subject and/or legally authorized representative unwilling to provide consent/assent for participation in the 15-year follow-up period, required if DARIC T cell therapy is administered
10. Presence of any condition that, in the opinion of the investigator, would prohibit the subject from undergoing treatment under this protocol
11. Considered by the investigator to be unable to tolerate a lymphodepleting regimen
12. Subject has a contraindication to receiving rapamycin

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2041-01-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events associated with SC-DARIC33 cell product infusions will be assessed | 28 days post-infusion
  The type, frequency, severity, and duration of adverse events will be summarized
Ability to successfully manufacture SC-DARIC33 | 28 days
  Measure of the number of successfully manufactured SC-DARIC33 products

SECONDARY OUTCOMES:
Acute Myeloid Leukemia response to SC-DARIC in subjects with relapsed or refractory CD33+ myeloid leukemia will be assessed | 28 days post-infusion
  The efficacy of the SC-DARIC33 assessed based on the bone marrow aspirate testing following SC-DARIC infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States